CLINICAL TRIAL: NCT05580328
Title: An Exploratory Clinical Study of Photodynamic Therapy With Hematoporphyrin Injection Combined With Sonodynamic Therapy in the Treatment of Inoperable Cholangiocarcinoma
Brief Title: An Exploratory Clinical Study of Photodynamic Therapy Combined With Sonodynamic Therapy in Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiaofeng Jiang, Professor, Second Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-YY-09
Record Dates: First submitted 2022-09-29; First posted 2022-10-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment group (Experimental): Hematoporphyrin injection is a new drug for tumor photodynamic therapy approved by the State Food and Drug Administration of China. It is a representative drug of domestic photosensitizer with independent intellectual property rights developed and produced by Chongqing Huading Modern Biological Pharmaceutical Co., Ltd.
  In the third phase clinical trial, the dosage of hematoporphyrin injection (5mg/kg) should be given intravenously 48-72 hours before laser irradiation for diagnosis and treatment, and skin test should be conducted before injection. Diagnostic laser wavelength is 514.5nm, power density is 10mW/cm2, therapeutic laser wavelength is 630-690nm, average output power density is 400mW/cm, and optical dose density is 200-400J/cm2 The chemical structure formula of hematoporphyrin is: C34H38N4O6, molecular weight: 598.70
  Interventions: Drug: Hematoporphyrin Injection actived by photodynamic therapy combined with Sonodynamic Therapy

INTERVENTIONS:
Drug: Hematoporphyrin Injection actived by photodynamic therapy combined with Sonodynamic Therapy — Hematoporphyrin in tumor tissue will be greatly enhanced by the combination of Sonodynamic Therapy and Photodynamic Therapy and achieve better treatment effect.

SUMMARY:
After enrollment, they received photodynamic therapy and sonodynamic therapy for a maximum of 2 times, and the longest treatment time was 6 months.The investigator will judge whether the second photodynamic therapy+ sonodynamic therapy treatment treatment is necessary according to the tolerance and tumor progress of the subject. The second photodynamic therapy+ sonodynamic therapy treatmentwill be carried out at the end of the sixth month. After the treatment period, the patients will be followed up once in the first, third and sixth months respectively, and then every three months. The observation and follow-up were carried out from the first subject after randomization to the end of 24 months after the last case.

The inspection and follow-up evaluation on the 7th day of the treatment period, including vital sign examination, blood routine examination, urine routine examination, blood biochemical examination, electrocardiogram examination, recording the number of times of plastic stent/metal stent drainage/drainage tube replacement, evaluation of physical status scale, evaluation of quality-of-life scale, recording concomitant medication and adverse events.

At the end of the first, third and sixth month, you need to come to the hospital for follow-up evaluation. In the test group, the investigator shall judge whether the second photodynamic therapy is needed at the end of the sixth month according to the tolerance and tumor progression of the subject. Before receiving the next photodynamic therapy, your body and quality of life must be evaluated according to KPS score and quality of life scale Arrange laboratory and relevant examinations. If the second photodynamic therapy is needed, continue to record the concomitant medication and adverse events at this stage.

During the follow-up period, after the longest treatment period of 6 months, a follow-up was conducted every 3 months until the end of 24 months after the last subject was enrolled in the scheme. Your survival, replacement of plastic stent/metal stent/drainage tube, biliary drainage, treatment methods for cholangiocarcinoma and serious adverse events were recorded during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, male or female
* Patients with advanced cholangiocarcinoma confirmed by imaging, biopsy or cytology (including hilar cholangiocarcinoma, middle and lower segment cholangiocarcinoma, ampullary tumor, etc.) who do not have the conditions for surgical resection due to vascular invasion and metastasis
* Karnofsky score ≥ 70
* The patient voluntarily participated in the trial and signed the informed consent form

Exclusion Criteria:

* The expected life span is less than 3 months
* White blood cells of subjects < 3.0 × 109/L, or hemoglobin is less than 80 g/L, or neutrophil is less than 1.5 × 109/L, or platelet<75 × 109/L, or other blood system diseases
* Blood creatinine > 1.5 times the upper limit of normal value
* In patients with severe liver function damage, ALT and/or AST>5 times the upper limit of normal value
* Have porphyria or allergy to porphyrin drugs
* Patients with active and untreated infection and/or acute bacterial or fungal infection (except biliary tract infection and cholecystitis) at the time of enrollment
* Severe hypertension (180mmhg / 110mmhg) that has not been controlled after intervention treatment, or serious complications of hypertension, or serious complications of diabetes
* Have serious heart, lung and central nervous system diseases
* Patients with mental illness or mental retardation who cannot correctly describe their feelings or cannot take medicine as instructed by the doctor
* Female patients who have become pregnant or may become pregnant and are unwilling to take reasonable and effective contraceptive measures, or are breastfeeding, or patients and/or sexual partners hope to become pregnant during the study period
* In addition to the above, the investigator determined that the patients were not suitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Size of tumor evaluated by CT | CT will be performed at the 24th months.
  Vealued by the size of tumor which was measured by CT